CLINICAL TRIAL: NCT00643240
Title: Phase I Open Label, Single Arm Escalation Trial to Evaluate the Biodistribution and Safety of BU-12 in Patients With Advanced Leukemia
Brief Title: Yttrium Y 90 Anti-CD19 Antibody BU-12 in Patients With Advanced Relapsed or Refractory Acute Lymphoblastic Leukemia or Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006LS057; MT2006-09 (Other: Blood and Marrow Transplantation Program); UMN-0611M96887 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-03-25; First posted 2008-03-26 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 111 In-BU-12 (Experimental): 111In-BU-12 is the 111Indium-labeled murine monoclonal antibody used for imaging and dosimetry.
  Interventions: Radiation: yttrium Y 90 anti-CD19 monoclonal antibody BU12; Radiation: 111In-BU-12

INTERVENTIONS:
Radiation: yttrium Y 90 anti-CD19 monoclonal antibody BU12 — Patients in whom the biodistribution is as expected (unaltered) AND a HAMA response does not develop will receive a single dose of 90Y-BU-12 in a dose escalated manner to establish the maximum tolerated dose (MTD) of 90Y-BU-12 over 60 minutes on Day 0. A single course of BU-12 includes the imaging dose of 111In-BU-12 followed 7-8 days later by the therapy dose of 90YBU- 12.
  Other Names: 90Y-BU-12
Radiation: 111In-BU-12 — Patients receive indium-111 BU-12 IV over 60 minutes on day 0
  Other Names: indium-111 BU-12

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can find cancer cells and carry cancer-killing substances to them without harming normal cells. This may be effective treatment for leukemia.

PURPOSE: This phase I trial is studying the best dose of yttrium Y 90-labeled monoclonal antibody BU-12 in treating patients with advanced relapsed or refractory acute lymphoblastic leukemia or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the biodistribution of indium-111 BU-12 in patients with refractory CD19+ leukemia.

Secondary

* To determine the maximum tolerated dose of yttrium Y 90 anti-CD19 antibody BU-12
* Determine the human anti-mouse antibody (HAMA) response.
* To define, preliminarily, the antitumor activity of yttrium Y 90 anti-CD19 antibody BU-12.

OUTLINE: Patients receive yttrium Y 90 anti-CD19 antibody BU-12/indium-111 BU-12 IV over 60 minutes on day 0 and undergo whole-body imaging on days 0, 1, 3, 4, and 7. Patients also undergo blood collection and bone marrow biopsy periodically for dosimetry calculations and pharmacokinetics.

After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD19-positive (> 25% by flow cytometry evaluation of bone marrow blasts) disease of 1 of the following types:

  * Primary refractory or relapsed acute lymphoblastic leukemia (ALL) defined as persistent disease following a minimum of two different standard effective chemotherapy induction attempts at time of diagnosis or at relapse
  * Chronic Lymphocytic leukemia (CLL) following blast crisis (≥15% bone marrow blasts following a minimum of one standard effective chemotherapy induction attempt)
* Human anti-mouse antibody (HAMA) must be negative
* Patients who have relapsed ≥ 60 days following an autologous or allogeneic transplant are eligible if all other eligibility criteria are met
* No active central nervous system (CNS) disease
* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy > 8 weeks
* Total bilirubin ≤ 2.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* LVEF ≥ 45% by MUGA/ECHO
* Oxygen saturation on room air > 92% and no oxygen requirement
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients mus use effective contraception

Exclusion criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to of yttrium Y 90 anti-CD19 antibody BU-12 or other agents used in study
* Uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive
* Active graft-vs-host disease
* Less than 4 weeks since prior agents and recovered
* Less than 7 days since prior therapy with any biologic agent, defined as a growth factor or cytokine
* Less than 3 months since prior antibody or biologic anticancer therapy (e.g., alemtuzumab or epratuzumab)
* Other concurrent investigational agents
* Patients with peripheral blasts > 5,000/uL may receive concurrent hydroxyurea

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Biodistribution of indium-111 BU-12 | Immediately post infusion, 4-6 hours after infusion and Days 1, 3, 4 and 7 after infusion
  Perform a whole body scan acquiring both anterior and posterior images at a speed of 10 cm/min (20 minute scan) using a medium energy collimator, a 256 x 1024 computer acquisition matrix and acquisition photo peak settings of 172 and 247 keV with 15% windows.

SECONDARY OUTCOMES:
Maximum tolerated dose of yttrium Y 90 anti-CD19 antibody BU-12 | Beginning Day 1 of treatment
  DLT will be defined as bone marrow aplasia > 6 weeks duration from the first treatment day; specifically, failure to recover peripheral ANC > 500/μL and platelets > 20,000/μL documented by bone marrow aplasia, not malignant infiltration - Any NCI CTCAE v 3.0 grade 3 non-hematologic toxicity except for allergic reactions to radiolabeled BU-12 will be dose limiting. If the BU-12 antibody is very allergenic, then ≥ grade 3 allergic reactions will be dose limiting.
Presence or absence of a human antibody to murine antibody | baseline, 28 and 60 days post therapy, and at 6 months post therapy
  Presence or absence of a human antibody to murine antibody at baseline, 28 and 60 days post therapy, and at 6 months post therapy
Number of Patients by Clinical Response | day 28 and day 60
  Patients evaluable for DLT will be assessed for response at day 28 and day 60 post therapy dose (event is whether or not the patient has a Complete Remission, Partial Remission, Stable Disease, Refractory Disease, Relapsed Disease). The proportion of patients by disease status will be reported.
Time to Clinical Response | Day 28, 60, 6 Months
  Time-to-event will be measured from date of therapy dose.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Weigel, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States